CLINICAL TRIAL: NCT06592014
Title: Repurposing Lithium as a Disease-modifying Therapy in Parkinson's Disease: an Open-label Extension Trial.
Brief Title: Lithium for Parkinson's: an Extension Trial
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Thomas Guttuso, Professor of Neurology, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008239
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
Keywords: lithium; biomarker; free water; neurofilament light chain
MeSH Terms: conditions — Parkinson Disease; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lithium aspartate (Experimental): Lithium aspartate with dosage adjusted to achieve a serum lithium level of 0.25-0.50mmol/L
  Interventions: Dietary Supplement: Lithium aspartate

INTERVENTIONS:
Dietary Supplement: Lithium aspartate — Lithium aspartate with dosage adjusted to serum lithium level 0.25-0.50mmol/L

SUMMARY:
This study will examine the effects of 24 weeks of lithium therapy achieving serum lithium levels of 0.25-0.50mmol/L on MRI and blood-based biomarkers in Parkinson's disease patients who have completed one of our current 24-week lithium clinical trials.

DETAILED DESCRIPTION:
In observational studies, small daily doses of lithium from smoking cigarettes have been associated with a 77% reduced risk of developing Parkinson's disease (PD). In addition, lithium therapy has been effective in preventing neuronal death and behavioral symptoms in several PD animal models. Recently, our group has shown 24-weeks of low-dose lithium therapy in PD to be associated with improvements in both MRI and blood-based biomarkers implying that lithium may be slowing the progression of the disease. However, these findings stemmed from only three of four patients receiving MRIs. Our group is now conducting two larger studies enrolling a total of 35 PD patients who are being treated with either 45mg/day or 20mg/day of lithium or placebo therapy for 24 weeks. Because our earlier study showed maximum improvements in PD biomarkers in patients with serum lithium levels of 0.25-0.50mmol/L and there are large interpatient variations in serum lithium levels achieved from the same lithium dosage, this present study will adjust lithium dosing in each patient to achieve this target serum lithium level for an additional 24 weeks. MRI and blood-based biomarker changes from Baseline will be compared in patients with serum lithium levels ≥ 0.25mmol/L and <0.25mmol/L from one of the 24-week studies and within individual patients. Results from this study may identify a target serum lithium level range associated with maximum improvements in PD biomarkers that can be used in the design of future, larger lithium PD lithium trials, which may eventually support lithium as a disease-modifying therapy for PD that could improve patients' long-term prognoses.

ELIGIBILITY:
1. All PD patients completing STUDY00007253 or STUDY00008239 at the University at Buffalo will be eligible.
2. No unstable cardiac, medical, neurologic or psychiatric condition in the opinion of the PI.
3. No current use of illicit drugs or current alcohol abuse in the opinion of the PI.
4. No history of brain surgery or possible need for brain surgery including deep brain stimulation (DBS) for at least 24 weeks in the opinion of the PI.
5. Women with child bearing potential will need a negative pregnancy test and not be nursing an infant at screening. Women with child bearing potential will need to report using barrier method or hormonal contraception.
6. Willing and able to sign informed consent and follow study procedures.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Free Water | 24 Weeks.
  Change in MRI-assessed free water in posterior substantia nigra, dorsomedial nucleus of the thalamus and nucleus basalts of Meynert.
Serum neurofilament light chain | 24 weeks
  Change in serum neurofilament light chain

SECONDARY OUTCOMES:
Peripheral blood mononuclear cell (PBMC) Nurr1 mRNA levels by real-time polymerase chain reaction (PCR) | 24 weeks
  Change in PBMC Nurr1
PBMC superoxide dismutase 1 (SOD-1) mRNA levels | 24 weeks
  Change in PBMC SOD-1
PBMC phosphorylated (p) and total (t) levels of pS9 and total-glycogen synthase kinase 3B (GSK-3B) | 24 weeks
  Change in PBMC pS9 and t-GSK-3B
PBMC pThr308, pS473 and t-protein kinase B (Akt) | 24 weeks
  Change in pThr308, pS473 and t-Akt
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part III | 24 weeks
  Change in MDS-UPDRS part III scores, Assessed in the "on" state. Score range 0-132 with higher scores indicating worse outcomes.
Parkinson's Anxiety Scale | 24 weeks
  Change in Parkinson's Anxiety Scale scores, Score range 0-48 with higher scores indicating worse outcomes.
Geriatric Depression Scale-15 | 24 weeks
  Change in Geriatric Depression Scale-15 scores, Score range 0-15 with higher scores indicating worse outcomes.
Fatigue Severity Scale | 24 weeks
  Change in Fatigue Severity Scale scores, Score range 9-63 with higher scores indicating worse outcomes.
Insomnia Severity Index | 24 weeks
  Change in Insomnia Severity Index, Score range 0-28 with higher scores indicating worse outcomes.
Parkinson's Disease Questionnaire-8 | 24 weeks
  Change in Parkinson's Disease Questionnaire-8 scores, Score range 0-32 with higher scores indicating worse outcomes.
Montreal Cognitive Assessment (MoCA) | 24 weeks
  Change in Montreal Cognitive Assessment (MoCA) version 1 and 2 scores, Score range 0-30 with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Guttuso, MD, Principal Investigator — University at Buffalo
Locations (1):
- UBMD Neurology, Williamsville, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient demographics and outcome measure results.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available after the study results are published.
Access Criteria: Researchers who have requested IPD from the PI.

REFERENCES:
- [Background] Guttuso T Jr, Shepherd R, Frick L, Feltri ML, Frerichs V, Ramanathan M, Zivadinov R, Bergsland N. Lithium's effects on therapeutic targets and MRI biomarkers in Parkinson's disease: A pilot clinical trial. IBRO Neurosci Rep. 2023 May 7;14:429-434. doi: 10.1016/j.ibneur.2023.05.001. eCollection 2023 Jun. PMID 37215748